CLINICAL TRIAL: NCT01855048
Title: A Randomized, Double-blind, Placebo-controlled, Clinical Study to Evaluate the Safety, Pharmacokinetics and Phyarmacodynamcs of a Single Intravenous Dose of N-Rephasin® SAL200, in Healthy Male Valunteers
Brief Title: A Study to Evaluate the Safety, Pharmacokinetics and Pharmacodynamics of N-Rephasin® SAL200 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Intron Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SAL200-1A
Record Dates: First submitted 2013-05-03; First posted 2013-05-16 (Estimated); Results first posted 2021-11-03 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-09

CONDITIONS: Healthy Volunteers; Anti-Bacterial Agents; Methicillin-Resistant Staphylococcus Aureus
Keywords: N-Rephasin® SAL200; endolysin; Placebo

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- N-Rephasin® SAL200 (Experimental): N-Rephasin® SAL200, 0.1 mg/kg, 0.3 mg/kg, 1 mg/kg, 3 mg/kg, 10 mg/kg
  Interventions: Biological: N-Rephasin® SAL200
- INT200-Placebo (Placebo Comparator): Placebo
  Interventions: Other: INT200-Placebo

INTERVENTIONS:
Biological: N-Rephasin® SAL200 — continuous intravenous infusion over 60 minutes
  Arms: N-Rephasin® SAL200
Other: INT200-Placebo — Formulation buffer for continuous intravenous infusion over 60 minutes
  Arms: INT200-Placebo

SUMMARY:
The Objectives of this study is to evaluate the safety, pharmacokinetics and pharmacodynamics of single dose of N-Rephasin® SAL200 in healthy male subjects.

DETAILED DESCRIPTION:
The purposes of this study are to evaluate the pharmacokinetics, and pharmacodynamics and safety of an experimental intravenous medication, N-Rephasin® SAL200 in healthy male. Participants will include 36 male volunteers. Participants will be grouped according to dosage of N-Rephasin® SAL200 including placebo (0 mg/kg). Study procedures include: check of vital signs, reporting any experienced side effects, physical examination including assessment of the cardiovascular system, and blood sample collection for monitoring of pharmacokinetics, pharmacodynamics and antibody production etc. Participants will be involved in study related procedures for up to 50 days after injection.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subject whose age is 20 ~ 45 at the time of screening visit.
* Body weight of ≥50kg and <90kg, while within ±20% of the ideal body weight. [ideal body weight(kg) = {height(cm)-100}x 0.9]
* Subject agreed to participate in the trial and to follow all of trial-related rules with a full understanding, after having a full account of the trial

Exclusion Criteria:

* Present disease(s) or medical history(ies) which is(are) clinically significant on liver, heart, nervous system, respiratory system, haemato-oncology, cardiovascular or psychopathy.
* Diagnosed or suspected infectious disease within 30 days in prior to the administration.
* Clinically significantly allergic to drug(s) containing AI of N-Rephasin® SAL200 or to other drugs including aspirin and antibiotics, or has medical history(ies) on such allergy.
* Already has taken other drug(s) containing AI of N-Rephasin® SAL200.
* Positive for Antibody of N-Rephasin® SAL200.
* SBP≤90mmHg or DBP≤50mmHg, otherwise, SBP≥150mmHg or DBP≥100mmHg in Vital sign which was measured after taking 3 minutes of resting in sitting position.
* Has medical history of drug abuse or positive to drug abuse in urine drug screening.
* Has taken any prescription drug(s) or herbal medicine(s) within 14 days prior to the administration, otherwise, any OTC(Over the counter) (s) or vitamin(s) within 7 days prior to the administration(However, can participate in the study if investigator makes a decision that the subject can participate regardless the drug taken).
* Has taken any other study drugs within 2 months prior to the administration.
* Has donated blood(whole blood donation or component transfusion) within (2 months or 1 month, respectively) in prior to the administration, otherwise, has received blood transfusion within 1 month in prior to the administration.
* Smoke at present or positive to metabolism of nicotine in urine test.
* Drink regularly(over 21 units/week, 1 unit= 10 g of pure alcohol), otherwise, is not able to interrupt drinking and smoking in study period.
* Investigator made a decision that the subject is not eligible based on results of laboratory test or other reason.
* Not agree with contraception for 60days after the administration, otherwise, notification of pregnancy in case of his partner is pregnant for 90 days after the administration.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2013-08-06 (Actual); Primary Completion 2014-02-07 (Actual); Study Completion 2014-02-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: In Jin Jang, M.D., Ph. D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Loessner MJ. Bacteriophage endolysins--current state of research and applications. Curr Opin Microbiol. 2005 Aug;8(4):480-7. doi: 10.1016/j.mib.2005.06.002. PMID 15979390
- [Result] Fischetti VA. Bacteriophage lysins as effective antibacterials. Curr Opin Microbiol. 2008 Oct;11(5):393-400. doi: 10.1016/j.mib.2008.09.012. Epub 2008 Oct 14. PMID 18824123
- [Result] Loeffler JM, Nelson D, Fischetti VA. Rapid killing of Streptococcus pneumoniae with a bacteriophage cell wall hydrolase. Science. 2001 Dec 7;294(5549):2170-2. doi: 10.1126/science.1066869. PMID 11739958
- [Result] Wu JA, Kusuma C, Mond JJ, Kokai-Kun JF. Lysostaphin disrupts Staphylococcus aureus and Staphylococcus epidermidis biofilms on artificial surfaces. Antimicrob Agents Chemother. 2003 Nov;47(11):3407-14. doi: 10.1128/AAC.47.11.3407-3414.2003. PMID 14576095
- [Result] Schellekens H. Immunogenicity of therapeutic proteins. Nephrol Dial Transplant. 2003 Jul;18(7):1257-9. doi: 10.1093/ndt/gfg164. No abstract available. PMID 12808158
- [Derived] Jun SY, Jang IJ, Yoon S, Jang K, Yu KS, Cho JY, Seong MW, Jung GM, Yoon SJ, Kang SH. Pharmacokinetics and Tolerance of the Phage Endolysin-Based Candidate Drug SAL200 after a Single Intravenous Administration among Healthy Volunteers. Antimicrob Agents Chemother. 2017 May 24;61(6):e02629-16. doi: 10.1128/AAC.02629-16. Print 2017 Jun. PMID 28348152
- See also: FDA, Guidance for Industry, Estimating the Maximum Safe Starting Dose inInitial Clinical Trials for Therapeutics in Adult Healthy Volunteers, 2005. — https://www.semanticscholar.org/paper/Guidance-for-Industry-Estimating-the-Maximum-Safe-Alert/8750b5d4c6564d44ac84826e3760f15ea0b836de

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment have completed in a single center (Seoul National University Hospital) from Nov. 2013 and the completion date is Feb. 2014.
Pre-assignment Details: 57 subjects were screened and 36 subjects met the eligibility criteria.
Groups:
- N-Rephasin® SAL200, 0.1mg/kg; N-Rephasin® SAL200, 0.3 mg/kg; N-Rephasin® SAL200, 1 mg/kg; N-Rephasin® SAL200, 3 mg/kg; N-Rephasin® SAL200, 10 mg/kg: N-Rephasin® SAL200: continuous intravenous infusion over 60 minutes
Period: Overall Study
Arm/Group | INT200-Placebo | N-Rephasin® SAL200, 0.1mg/kg | N-Rephasin® SAL200, 0.3 mg/kg | N-Rephasin® SAL200, 1 mg/kg | N-Rephasin® SAL200, 3 mg/kg | N-Rephasin® SAL200, 10 mg/kg
Started | 9 | 3 | 6 | 6 | 6 | 6
Completed | 9 | 2 | 6 | 6 | 5 | 6
Not Completed | 0 | 1 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: one subject in the 1 mg/kg dose group was 171.3 cm in height and weighed 81 kg at the screening, indicating that this subject was not within the range of ideal body weight (51.3-77.0 kg) for the subject's height, but the subject was enrolled in the study. The investigators judged that that subject was not at increased risk of adverse events in comparison with other subjects. Subject completed the remaining study procedures as scheduled in the study protocol without showing adverse events.
Groups:
- N-Rephasin® SAL200 0.1(mg/kg): N-Rephasin® SAL200, 0.1 mg/kg
  N-Rephasin® SAL200: continuous intravenous infusion over 60 minutes
- N-Rephasin® SAL200 0.3(mg/kg): N-Rephasin® SAL200, 0.3 mg/kg
  N-Rephasin® SAL200: continuous intravenous infusion over 60 minutes
- N-Rephasin® SAL200 1(mg/kg): N-Rephasin® SAL200,
  1 mg/kg
  N-Rephasin® SAL200: continuous intravenous infusion over 60 minutes
- N-Rephasin® SAL200 3(mg/kg): N-Rephasin® SAL200, 3 mg/kg
  N-Rephasin® SAL200: continuous intravenous infusion over 60 minutes
- N-Rephasin® SAL200 10(mg/kg): N-Rephasin® SAL200, 10 mg/kg
  N-Rephasin® SAL200: continuous intravenous infusion over 60 minutes
- Total: Total of all reporting groups
Arm/Group | N-Rephasin® SAL200 0.1(mg/kg) | N-Rephasin® SAL200 0.3(mg/kg) | N-Rephasin® SAL200 1(mg/kg) | N-Rephasin® SAL200 3(mg/kg) | N-Rephasin® SAL200 10(mg/kg) | INT200-Placebo | Total
Number analyzed (Participants) | 3 | 6 | 6 | 6 | 6 | 9 | 36
Age, Customized [Mean (Full Range); unit: Years] | 25.3 [25 to 26] | 27.8 [23 to 33] | 29.8 [23 to 39] | 23.7 [20 to 27] | 30.5 [24 to 38] | 26.2 [22 to 29] | 27.4 [20 to 39]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 3 | 6 | 6 | 6 | 6 | 9 | 36
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 3 | 6 | 6 | 6 | 6 | 9 | 36
Region of Enrollment [Number; unit: participants]
  South Korea | 3 | 6 | 6 | 6 | 6 | 9 | 36
Body weight [Mean (Full Range); unit: kg] | 67.1 [64.1 to 72.2] | 65.5 [54.9 to 76.2] | 74.0 [67.6 to 80.5] | 69.1 [58.7 to 78.8] | 68.7 [64.0 to 72.4] | 68.1 [63.1 to 73.5] | 68.9 [54.9 to 80.5]
Height [Mean (Full Range); unit: cm] | 176.8 [171.2 to 181.2] | 171.3 [165.2 to 175.9] | 175.1 [171.3 to 179.8] | 174.8 [171.3 to 177.3] | 170.5 [163.7 to 178.6] | 174.5 [169.8 to 179.3] | 173.6 [163.7 to 181.2]

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of the Safety of N-Rephasin® SAL200 in Healthy Human Volunteers
Time Frame: Up to 50 days after administration
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: INT200-Placebo, IV administration
- N-Rephasin® SAL200 (0.1 mg/kg): Study drug 0.0056 mL/kg, IV administration
- N-Rephasin® SAL200 (0.3 mg/kg): Study drug 0.017 mL/kg, IV administration
- N-Rephasin® SAL200 (1 mg/kg): Study drug 0.056 mL/kg, IV administration
- N-Rephasin® SAL200 (3 mg/kg): Study drug 0.167 mL/kg, IV administration
- N-Rephasin® SAL200 (10 mg/kg): Study drug 0.556 mL/kg, IV administration
Arm/Group | Placebo | N-Rephasin® SAL200 (0.1 mg/kg) | N-Rephasin® SAL200 (0.3 mg/kg) | N-Rephasin® SAL200 (1 mg/kg) | N-Rephasin® SAL200 (3 mg/kg) | N-Rephasin® SAL200 (10 mg/kg)
Number analyzed (Participants) | 9 | 3 | 6 | 6 | 6 | 6
Participants
  Number of Subjects with at least one AE | 1 | 0 | 2 | 1 | 2 | 6
  Number of Subjects with at least one drug-related AE | 1 | 0 | 2 | 1 | 0 | 6

2. Other Pre Specified Outcome: Pharmacokinetic Parameters After Single IV Administration of N-Rephasin® SAL200 [Effective t1/2 (h)]
Time Frame: 0, 4, 8, 12, 16, 20, 24 hours post-dose
Measure: Mean (Standard Deviation); unit: h
Groups:
- N-Rephasin® SAL200 0.1mg/kg: Study drug 0.0056 mL/kg, IV administration
- N-Rephasin® SAL200 0.3mg/kg: Study drug 0.017 mL/kg, IV administration
- N-Rephasin® SAL200 1mg/kg: Study drug 0.056 mL/kg, IV administration
- N-Rephasin® SAL200 3mg/kg: Study drug 0.167 mL/kg, IV administration
- N-Rephasin® SAL200 10mg/kg: Study drug 0.556 mL/kg, IV administration
Arm/Group | N-Rephasin® SAL200 0.1mg/kg | N-Rephasin® SAL200 0.3mg/kg | N-Rephasin® SAL200 1mg/kg | N-Rephasin® SAL200 3mg/kg | N-Rephasin® SAL200 10mg/kg
Number analyzed (Participants) | 3 | 6 | 6 | 6 | 6
h | 0.04 (0.02) | 0.04 (0.01) | 0.25 (0.05) | 0.38 (0.06) | 0.38 (0.05)

3. Other Pre Specified Outcome: Pharmacodynamics Evaluation of N-Rephasin® SAL200 : Mean Concentration of Bactericidal Activity After Single Dose of N-Rephsin® SAL200 IV Administration
Time Frame: up to 2hours
Measure: Mean (Standard Deviation); unit: μg/mL
Groups:
- N-Rephasin® SAL200 0.1 mg/kg: Study drug 0.0056 mL/kg, IV administration
- N-Rephasin® SAL200 0.3 mg/kg: Study drug 0.017 mL/kg, IV administration
- N-Rephasin® SAL200 1 mg/kg: Study drug 0.056 mL/kg, IV administration
- N-Rephasin® SAL200 3 mg/kg: Study drug 0.167 mL/kg, IV administration
- N-Rephasin® SAL200 10 mg/kg: Study drug 0.556 mL/kg, IV administration
Arm/Group | N-Rephasin® SAL200 0.1 mg/kg | N-Rephasin® SAL200 0.3 mg/kg | N-Rephasin® SAL200 1 mg/kg | N-Rephasin® SAL200 3 mg/kg | N-Rephasin® SAL200 10 mg/kg
Number analyzed (Participants) | 3 | 6 | 6 | 6 | 6
μg/mL
  0h | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  1h | 0 (0) | 0 (0) | 0.13 (0.05) | 0.22 (0.10) | 0.40 (0.13)
  1.5h | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0.15 (0.06)
  2h | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0.04 (0.05)

4. Other Pre Specified Outcome: Pharmacokinetic Evaluation of N-Rephasin® SAL200 at the Administered Doses by Analysis of Concentration of N-Rephasin® SAL200 in Serum [Cmax (µg/ml)]
Time Frame: Day 1 to 2
Measure: Mean (Standard Deviation); unit: µg/ml
Arm/Group | N-Rephasin® SAL200 0.1mg/kg | N-Rephasin® SAL200 0.3mg/kg | N-Rephasin® SAL200 1mg/kg | N-Rephasin® SAL200 3mg/kg | N-Rephasin® SAL200 10mg/kg
Number analyzed (Participants) | 3 | 6 | 6 | 6 | 6
µg/ml | 0.04 (0.01) | 0.09 (0.04) | 0.82 (0.50) | 7.10 (5.39) | 55.99 (10.37)

5. Other Pre Specified Outcome: Pharmacokinetic Evaluation of N-Rephasin® SAL200 at the Administered Doses by Analysis of Concentration of N-Rephasin® SAL200 in Serum [Cmax/D (µg/ml/mg)]
Time Frame: Day 1 to 2
Measure: Mean (Standard Deviation); unit: µg/ml/mg
Arm/Group | N-Rephasin® SAL200 0.1mg/kg | N-Rephasin® SAL200 0.3mg/kg | N-Rephasin® SAL200 1mg/kg | N-Rephasin® SAL200 3mg/kg | N-Rephasin® SAL200 10mg/kg
Number analyzed (Participants) | 3 | 6 | 6 | 6 | 6
µg/ml/mg | 0.01 (0.001) | 0.005 (0.001) | 0.01 (0.01) | 0.03 (0.02) | 0.08 (0.01)

6. Other Pre Specified Outcome: Pharmacokinetic Evaluation of N-Rephasin® SAL200 at the Administered Doses by Analysis of Concentration of N-Rephasin® SAL200 in Serum [AUC Last (µg*h/ml)]
Time Frame: Day 1 to 2
Measure: Mean (Standard Deviation); unit: µg*h/ml
Arm/Group | N-Rephasin® SAL200 0.1mg/kg | N-Rephasin® SAL200 0.3mg/kg | N-Rephasin® SAL200 1mg/kg | N-Rephasin® SAL200 3mg/kg | N-Rephasin® SAL200 10mg/kg
Number analyzed (Participants) | 3 | 69 | 6 | 6 | 6
µg*h/ml | 0.03 (0.005) | 0.05 (0.02) | 0.57 (0.31) | 7.26 (3.42) | 59.79 (9.03)

ADVERSE EVENTS:
Time Frame: Up to 50 Days ± 7 Days
Arm/Group | INT200-Placebo | N-Rephasin® SAL200, 0.1mg/kg | N-Rephasin® SAL200, 0.3 mg/kg | N-Rephasin® SAL200, 1 mg/kg | N-Rephasin® SAL200, 3 mg/kg | N-Rephasin® SAL200, 10 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/3 | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/3 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 1/9 | 0/3 | 2/6 | 1/6 | 2/6 | 6/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | INT200-Placebo (N=9) | N-Rephasin® SAL200, 0.1mg/kg (N=3) | N-Rephasin® SAL200, 0.3 mg/kg (N=6) | N-Rephasin® SAL200, 1 mg/kg (N=6) | N-Rephasin® SAL200, 3 mg/kg (N=6) | N-Rephasin® SAL200, 10 mg/kg (N=6)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) — General disorders and administration site conditions
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — General disorders and administration site conditions
Rigors (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 4 (4) — General disorders and administration site conditions
Coughing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4)
Headache (Nervous system disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes